CLINICAL TRIAL: NCT03945461
Title: Return of Bowel Function After One or Two Level Anterior Lumbar Interbody Fusion With Chewing Gum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Maziyar A. Kalani, Consultant Neurosurgeon, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18-011849
Record Dates: First submitted 2019-04-04; First posted 2019-05-10 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Spondylosis; Spondylolisthesis; Neurogenic Claudication; Foraminal Stenosis
MeSH Terms: conditions — Spondylosis; Spondylolisthesis | interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gum chewing (Experimental): Chew xylitol based, peppermint flavored gum for 30 minutes every two hours during the hours of 7 am to 9 pm, for the first 24 hours after your surgery
  Interventions: Other: Chewing gum
- Standard Care (No Intervention): Standard hospital management with no deviations from usual care

INTERVENTIONS:
Other: Chewing gum — xylitol based, peppermint flavored gum
  Arms: Gum chewing

SUMMARY:
Researchers are trying to identify is chewing gum improves bowel function after anterior lumbar interbody fusion

DETAILED DESCRIPTION:
Aims, purpose, or objectives:

1. Observe changes in bowel pattern based on gum-chewing
2. Examine bowel function after anterior lumbar interbody fusion
3. Measure length of time to return of bowel function after anterior lumbar interbody fusion
4. Compare return of bowel function in patients who chew gum and patients standardized to usual post-operative care
5. Measure the hospital length of stay amongst study groups
6. Measure post-operative pain amongst study groups

Background (Include relevant experience, gaps in current knowledge, preliminary data, etc.):

One or two level anterior lumbar interbody fusions are designed to correct lumbar spondylosis and spondylolisthesis, which can cause debilitating back and leg pain. This surgery involves an anterior approach, which often requires displacement of bowel for the length of the surgery. Patients frequently have a slow return of bowel function secondary to anesthetic time, opioid use, and primarily due to the bowel displacement intraoperatively. Because this is a one or two level surgery, many patients would benefit from same-day discharge but often remain inpatient several days due to slow return of bowel function.

Gum chewing has been shown to decrease the time for return to bowel function (RBF) in colorectal and gynecology patients postoperatively.

Gum chewing and RBF has been studied in the spine population for posterior operations but not anterior spine surgery. This study aims to identify whether chewing gum has an impact on patient's report of pain, RBF, length of stay, and subjective report of satisfaction post-operatively. This could be an outpatient operation; however, pain and RBF often prevent patients from discharging home the same day of surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing one or two level anterior lumbar interbody fusion
2. Diagnosis of spondylosis, spondylolisthesis, revision of foraminal stenosis or neurogenic claudication

Exclusion Criteria:

1. Previous bowel surgery
2. Diagnosis of an inflammatory bowel disease
3. Allergy to xylitol
4. Pregnancy

Some participants may subsequently undergo a posterior spinal fusion on the same-day of surgery. They will not be excluded, but the investigators will include this group in a different data subset.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in bowel pattern based on gum-chewing | 24 hours after surgery
  Number of hours until return of bowel sounds

SECONDARY OUTCOMES:
Bowel function | Number of hours from admission to discharge up to 48 hours
  Number of hours until return of flatus
Length of time to return of bowel function after anterior lumbar interbody fusion | Number of hours from admission to discharge up to 48 hours
  Number of hours until complete bowel movement
Total length of hospital | Number of hours from admission to discharge up to 48 hours
  Number of hours of hospital stay
Pain score | 24 hours post-operatively
  On a scale of 0 (zero pain) and 10 (worst pain)

CONTACTS AND LOCATIONS:
Overall Officials: Maziyar Kalani, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials